CLINICAL TRIAL: NCT04115254
Title: A Master Protocol of Stereotactic Magnetic Resonance Guided Adaptive Radiation Therapy (SMART)
Brief Title: Stereotactic Magnetic Resonance Guided Radiation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jonathan Leeman, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-353
Record Dates: First submitted 2019-09-26; First posted 2019-10-03 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Pancreas Cancer; Lung Cancer; Renal Cancer; Adrenal Metastases; Prostate Cancer; Liver Metastases; Oligoprogressive Nodal Metastases; Metachronous Nodal Metastases; Synchronous Nodal Metastases; Mesothelioma; Spine Metastases; Brain Metastases; Borderline Resectable Pancreatic Carcinoma
Keywords: Magnetic Resonance Imaging (MRI); MRIdian Linear Accelerator; Pancreas Cancer; Lung Cancer; Renal Cancer; Adrenal Metastases; Prostate Cancer; Liver Metastases; Oligoprogressive; Metachronous; Synchronous; Spine; Prostate Boost; Pelvic Re Irradiation
MeSH Terms: conditions — Pancreatic Neoplasms; Lung Neoplasms; Kidney Neoplasms; Prostatic Neoplasms; Mesothelioma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: All participants will be assigned to one treatment arm only depending on their cancer type, and will be taken off study once treatment and follow up are complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (19):
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Pancreatic (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Renal (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Central Lung (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Adrenal Metastases (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Liver Metastases (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Metachronous Oligometastatic Nodes (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Oligoprogressive Oligometastatic Nodes/Soft Tissue (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Synchronous Oligometastatic Nodes/Soft Tissue (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Prostate (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Borderline Resectable Pancreas (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Brain Metastases (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Mesothelioma (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Prostate Boost (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Pelvic Re-Irradiation (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Spine (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Single-Fraction Kidney Tumors (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--1/3 Fraction for Oligometastatases in the Abdomen/Pelvis (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Post-Operative Radiation Therapy in Lung Cancer (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac
- PHASE 1: SBRT MR IMAGE GUIDANCE/ADAPTATION--Mediastinal and Hilar Lymph Nodes (Experimental): SMART will be administered per each individual disease site standards
  Interventions: Radiation: MR-guided Linac

INTERVENTIONS:
Radiation: MR-guided Linac — Radiation will be delivered on an MR-guided Linear Accelerator

SUMMARY:
This is a master prospective Phase I-II trial evaluating feasibility and efficacy of stereotactic magnetic resonance (MR) guided adaptive radiation therapy (SMART) in patients with cancer.

* The phase 1 study will evaluate the feasibility and safety of delivering SMART in patients with cancer.
* Phase 2 will evaluate efficacy of SMART with specific reference to tumor control and improvement in patient reported outcome measures

DETAILED DESCRIPTION:
This research study is a feasibility study, which means it is the first-time investigators at this institution are examining this type of MR-guided radiation to treat cancer.

The U.S. Food and Drug Administration (FDA) has approved this device as a treatment option for cancer.

In this research study, the investigators are hoping to determine if adjusting radiation treatments based on daily MRI has a feasible way to deliver radiation for participants with pancreatic, lung or renal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed malignancy requiring stereotactic body radiation therapy. See specific disease site cohorts for more details.
* Tumor size ≤ 7cm
* Age 18 years of older.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Ability to understand and the willingness to sign a written informed consent document.
* Specific eligibility requirements for each disease site with be covered in each specific cohort.

Exclusion Criteria:

* Specific exclusion requirements for each disease site with be covered in each specific cohort
* History of allergic reactions attributed to gadolinium-based IV contrast.

  -- Note: If a patient will not receive contrast, this is not applicable
* Pregnant women are excluded from this study.
* Severe claustrophobia or anxiety
* Participants who cannot undergo an MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Delivery Success Rate for SMART across multiple tumors-Phase I | 1 year
  Enrolling patients and delivering SMART on the MR Linac
Tumor visualization-Phase I | 1 Year
  Assessing tumor using MR guidance before, during and after MR-guided treatment patient
Plan creation-Phase I | 1 Year
  Generating adaptive plans
Rate of Improvement in Tumor Control-Phase II | 1 Year
  Statistical power will be defined in each cohort individually and will be specific to each disease site tested.

SECONDARY OUTCOMES:
Number of Patients with Acute Toxicity-Phase I | 90 Days
  Any related ≥ Grade 3 AE which is possibly, probably or definitely related to SMART
Duration of treatment-Phase 1 | 90 Days
  Duration of treatment with goal of >80% of cases treated within 90 minutes
Number of treatment fractions-Phase1 | 90 Days
  Number of treatment fractions that would have resulted in unacceptably high dose (exceeding constraint) to an OAR without SMART
Number of Participants with long term toxicity-Phase II | 365 Days
  assessing long-term (12 month) toxicity in patients receiving SMART
Disease Specific Survival Rate-Phase II | 365 Days
  Kaplan-Meier curve estimates
Overall Survival Rate-Phase II | 365
  Kaplan-Meier curve estimates

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Leeman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Dr. Jonathan Leeman (jonathane_leeman@dfci.harvard.edu). The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BWH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Leeman JE, Shin KY, Droznin A, Catalano P, Cagney DN, Singer L, Oniyangi RD, Zhai K, Benham G, Chirmade S, Campbell J, Boyle S, Saranteas A, Williams CL, Huynh E, Han Z, Sudhyadhom A, Hu YH, Ferguson D, Singhrao K, Hsu SH, Bredfeldt J, Martin NE, Mancias JD, Mamon HJ, Van Dams R, Venkatachalam V, Tanguturi SK, Huynh MA, Fitzgerald KJ, Elhalawani H, Bitterman DS, Schoenfeld JD, Nguyen P, Haas-Kogan DA, Mak R. Stereotactic magnetic resonance imaging-guided adaptive radiotherapy: a pooled analysis of a master prospective trial. J Natl Cancer Inst. 2025 Nov 1;117(11):2289-2297. doi: 10.1093/jnci/djaf208. PMID 40794880